CLINICAL TRIAL: NCT01828307
Title: Exercise: Addressing Stress in Relapse Prevention for Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: VA St. Louis Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeremiah Weinstock, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA033411-01A1 (NIH); 23298 (Other: Saint Louis University Institutional Review Board)
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Aftercare Treatment (Active Comparator): Standard aftercare treatment consists of once per week group counseling for six months. Aftercare includes the following topics: substance use, high-risk situations, coping and life skills training, focus groups for depression and anxiety, and AIDS education.
  Interventions: Behavioral: Standard Aftercare Treatment
- Standard Aftercare Treatment + Exercise Intervention (Experimental): In addition to attending standard aftercare treatment, participants will receive three 50-minute motivational enhancement therapy sessions focused on exercise, plus 24 weekly contingency management sessions for exercise.
  Interventions: Behavioral: Motivational enhancement therapy (MET); Behavioral: Contingency management; Behavioral: Standard Aftercare Treatment

INTERVENTIONS:
Behavioral: Motivational enhancement therapy (MET) — MET is a client-centered, directive method of enhancing intrinsic motivation for change by exploring and resolving ambivalence. In this intervention MET will focus on exercise.
  Arms: Standard Aftercare Treatment + Exercise Intervention
Behavioral: Contingency management — Contingency management is a behavioral treatment that utilizes extrinsic motivation by offering individuals tangible rewards such as prizes for completion of specific target behaviors. The target behavior in this study is exercise.
  Arms: Standard Aftercare Treatment + Exercise Intervention
Behavioral: Standard Aftercare Treatment — Aftercare includes the following topics: substance use, high-risk situations, coping and life skills training, focus groups for depression and anxiety, and AIDS education.

SUMMARY:
Relapse contributes significantly to the chronicity of substance use disorders, one of the most costly medical/mental health problems facing our nation. The incorporation of exercise into relapse prevention efforts will address stress, a critical factor in relapse, provide other health benefits, and improve overall quality of life. Combined, these changes will reduce the risk of relapse to substance use while also lessening the burden of this psychiatric disorder upon society

DETAILED DESCRIPTION:
About half of all individuals who receive treatment for substance use disorders (SUD) relapse within a year. Stress and an individual's biological response to it are significant predictors of relapse. Thus, interventions that decrease stress and normalize an individual's biological response to stress are desperately needed. Exercise decreases stress and improves the body's regulation of stress. The proposed project will utilize exercise as a novel relapse prevention intervention with individuals who have recently completed inpatient SUD treatment. This project will evaluate the efficacy of a motivational intervention for exercise in a randomized clinical trial of 150 SUD patients beginning Aftercare treatment at the VA St. Louis Health Care System. Participants will be randomized to one of two interventions: (1) standard care (SC), or (2) standard care plus a motivational intervention targeting exercise that lasts for six months. Participants are followed every three months for one year. Results from this study will advance exercise as a new strategy for enhancing stress regulation and prevention of relapse in SUD populations.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing residential substance use disorders treatment at VA St. Louis Healthcare System
* Age 18 or older
* English speaking;
* Substance dependence
* Recent substance use
* Does not have high blood pressure
* Documented physician clearance to undergo exercise testing & exercise
* Plans to begin Aftercare at the clinic within the next two weeks

Exclusion Criteria:

* Severely disruptive behavior
* Serious uncontrolled psychiatric disorder
* Medical history in the past 6 months that contraindicates exercise
* Pregnancy, plans to get pregnant in the next six months.
* Currently breastfeeding
* Obese - class II
* Currently taking corticosteroids or hormonal contraceptives
* In recovery for pathological gambling
* Opiate dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2013-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in substance use (relapse) | At baseline and every three months for one year.
  Relapse is assessed during the duration of the study and is a time to event variable so it will be assess over time. Relapse is defined as drinking alcohol in excess of the National Institute on Alcohol Abuse and Alcohol (NIAAA) at-risk guidelines.
Change in moderate to vigorous physical activity | At baseline and every three months for one year.
  Moderate to vigorous physical activity frequency, duration and intensity will be assessed over time to examine changes in response to the intervention. Frequency is defined as how often and individual engages in moderate to vigorous physical activity. Duration is the amount of time (minutes) per episode that individual engages in moderate to vigorous physical activity. Intensity is defined two ways: (1) self-report rating of intensity and (2) metabolic equivalent of the moderate to vigorous physical activity.

SECONDARY OUTCOMES:
Change in stress reactivity over time. | At baseline and two additional times over one year.
  Stress reactivity is assess via a standardized psychosocial stressor paradigm that induces stress. Stress is assessed via salivary cortisol and self-report of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Weinstock, PhD, Principal Investigator — St. Louis University
Locations (1):
- VA St. Louis Health Care System - Jefferson Barracks Division, St Louis, Missouri, United States